CLINICAL TRIAL: NCT05075382
Title: Fracture and Neurological Injury: Prospective Multicentre Study on Risk Factors of Complications and Opioid Intake in Elbow Trauma
Brief Title: Fracture and Neurological Injury
Acronym: FIRE
Status: Withdrawn | Type: Observational
Why Stopped: A new version of the study will be submitted
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Dominique Rouleau, Principal investigator, Université de Montréal
Other Study IDs: FIRE
Record Dates: First submitted 2021-09-09; First posted 2021-10-12 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Elbow Fracture; Neurologic Deficits
Keywords: heterotopic ossification; traumatic brain injury
MeSH Terms: conditions — Elbow Fractures; Neurologic Manifestations; Ossification, Heterotopic; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Inflammatory factors (biomarkers, cytokines, chemokine such as interleukins, P substance, TNF alpha, osteopontin, S100B, NSE, GFAP)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pilot group: Group of 40 patients that will act as observationnal group for this study
  Interventions: Procedure: Elbow surgery for fracture

INTERVENTIONS:
Procedure: Elbow surgery for fracture — This group will undergo a surgery in order to fix a broken elbow.

SUMMARY:
The goal of the project is to describe novel factors affecting outcome after elbow fracture surgery with an in-depth evaluation of the role played by neuro inflammation from concomitant peripheral nerve injury or head injury in elbow fracture outcomes.

Among all upper limb fractures, elbow trauma is the most frequently associated with a severe impact on patient function and quality of life. One of the main reasons for poor outcomes is the complexity of the elbow joint, which involves three bones and two planes of motion, essential to position the hand in space. The flexion extension axis is crucial for eating and hygiene, while forearm pro-supination is mandatory for most professions, from office work to manual labour.

DETAILED DESCRIPTION:
Elbow fractures are a challenging clinical problem. The advancement of science and technology has made major contributions to improve outcomes. Nonetheless, even with an anatomical restoration of the bone architecture, many patients stay with major limitations and pain. In clinical practice, it is striking to see how two patients with a similar elbow injury can exhibit completely opposite presentations: one who has completely healed from his/her injury and the other who has a stiff and painful elbow. The reasons for these changeable outcomes are unclear.

The investigator hypothesize that many of the answers will be related to the neurological system. This would explain why most studies strictly focusing on the orthopedic component of upper limb injury have yielded little improvement in preventing the adverse outcomes experienced by patients.

Following surgical treatment of an elbow fracture, patients often present with complications. Indeed, one third of patients complain of ulnar nerve symptoms after distal humerus fracture fixation, and 50% of patients treated surgically for elbow fracture-dislocations will have disabling stiffness and heterotopic ossification (HO). HO results from resident cells of mesenchymal origin in soft tissues transforming into bone. Furthermore, approximately half of all patients with fractures feel significant pain leading to persistent narcotic intake 3 months post injury; 40% will suffer from a neuropathic type of pain, which is poorly controlled by narcotic medication. Opioid usage is also related to increased sensitivity to pain (hyperalgesia) and dissatisfaction. Complications from opioids prolonged usage are numerous, from constipation to death due to an overdose. Canada is second worldwide, behind the United States, when it comes to opioid use and mortality secondary to opioid use. The majority of opioid dependant users were first exposed to these substances through medical prescriptions. This makes it imperative to improve the scinetific community understanding of pain mechanisms and find alternative treatments to opiates in the management of these injuries.

In view of these observations, the investigator's research must focus on something other than "satisfactory radiological results" in patients with elbow injuries. To this end, a multidisciplinary approach is needed. The investigators oversee research in elbow trauma, neurotrauma and have an expertise in upper limb evaluation. To improve the understanding of the underlying physiological principles that contribute to pain and chronic stiffness, one of the topics targeted by the investigator is the role of neuro-inflammation (NI) in chronic pain and functional limitation in elbow trauma. The surgical factors that increase NI will allow surgeons to choose different therapeutic options and develop novel treatments.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years or older with an acute elbow fracture and dislocation less than a week old
* Open or arthroscopic surgery as the chosen treatment

Exclusion Criteria:

* Patient with a history of ipsilateral trauma, neurological disorder or major pathology.
* Patient unable to answer questionnaires.
* Patient unavailable for a one-year follow-up, for example from another country.
* Patient with vascular injury or open fracture
* Patient with a historic of TBI
* Patient with chronic medicated pain

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients presenting with elbow fracture that needs to be treated surgically.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of inflammatory factors with blood tests | Pre-op
  interleukins, P substance, TNF alpha, osteopontin, S100B, NSE, GFAP
Measurement of inflammatory factors with blood tests | During surgery
  interleukins, P substance, TNF alpha, osteopontin, S100B, NSE, GFAP
Measurement of inflammatory factors with blood tests | 3 months post-op
  interleukins, P substance, TNF alpha, osteopontin, S100B, NSE, GFAP

SECONDARY OUTCOMES:
Quick-DASH | Baseline, 2 weeks post-op, 3-6-12 months post-op
  Quick-DASH outcome measures (scores range from 0 (no disability) to 100 (most severe disability))
Patient rated elbow evaluation (PREE) | Baseline, 2 weeks post-op, 3-6-12 months post-op
  20 item questionnaire allowing patients to rate their levels of elbow pain and disability from 0 to 100 (0= no disability)
Range of motion | Baseline, 2 weeks post-op, 3-6-12 months post-op
  Evaluation of the elbow range of motion with goniometer by a train physical therapist
McGill Pain Questionnaire (MPQ-Short Form V2) | Baseline, 2 weeks post-op, 3-6-12 months post-op
  Self-reported measure of pain. No scale
Neuropathic pain questionnaire (SLANSS) | Baseline, 2 weeks post-op, 3-6-12 months post-op
  questionnaire designed to identify pain of predominantly neuropathic origin. A score over 12 signals a predominantly neuropathic type of pain
Euro-Qol Group 5Q5D | Baseline, 2 weeks post-op, 3-6-12 months post-op
  Questionnaire evaluating qaulity of life. No scale
Tourniquet | Per-op
  Verify our capacity to identify whether the use of tourniquet has an impact on neuroinflammation
Nerve dissection | Pero-op
  Verify our capacity to identify whether the nerve dissection has an impact on neuroinflammation

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Rouleau, MD, Principal Investigator — Université de Montréal

IPD SHARING:
Plan to Share IPD: No